CLINICAL TRIAL: NCT00624091
Title: Rationale, Design and Methods for the Early Surgery in Infective Endocarditis Study: a Multicenter, Prospective, Randomized Trial Comparing the State-of-the-Art Therapeutic Strategy Versus Early Surgery Strategy in Infective Endocarditis
Brief Title: Rationale, Design and Methods for the Early Surgery in Infective Endocarditis Study (ENDOVAL)
Acronym: ENDOVAL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Ciencias del Corazon (Other)
Responsible Party: Jose Alberto San Román Calvar, ICICOR
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDOVAL-1
Record Dates: First submitted 2008-02-02; First posted 2008-02-26 (Estimated); Last update posted 2008-02-26 (Estimated); Status verified 2008-02

CONDITIONS: Infective Endocarditis
Keywords: Early-surgery, infective endocarditis, in-hospital mortality
MeSH Terms: conditions — Endocarditis | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Early-surgery, within 48 hours from randomization
  Interventions: Procedure: Cardiac surgery
- 2 (Active Comparator): State-to-the-art group. Antibiotic treatment and surgery if emergency or sequelae of endocarditis as recommended in the guidelines
  Interventions: Procedure: State-to-the-art treatment

INTERVENTIONS:
Procedure: Cardiac surgery — Cardiac surgery within 48 hours of randomization
  Arms: 1
Procedure: State-to-the-art treatment — Antibiotic treatment and surgery if emergency or sequelae of endocarditis as recommended in the guidelines
  Arms: 2

SUMMARY:
Background: Prognosis of infective endocarditis is poor and has remained steady over the last four decades. Several nonrandomized studies suggest that early surgery could improve prognosis.

Methods: The early surgery in infective endocarditis study (ENDOVAL 1) is a multicenter, prospective, randomized study designed to compare the state-of-the-art therapeutic strategy (that advised by the international societies in their guidelines) with the early surgery strategy in high-risk patients with infective endocarditis. Patients with infective endocarditis without indication for surgery will be included if they meet at least one of the following: 1) early-onset prosthetic endocarditis; 2) Staphylococcus aureus endocarditis; 3) periannular complications; 4) new-onset conduction abnormalities; 5) vegetations longer than 10 mm in diameter; 6) new-onset severe valvular disfunction. A total of 216 patients will be randomized to either of the two strategies. Stratification will be done within 3 days of admission. In the early surgery arm, the procedure will be performed within 48 hours of randomization. The only event to be considered will be death within 30 days. The study will be extended to 1 year. In the follow-up substudy, death and a new episode of endocarditis will be regarded as events.

Conclusion: The early surgery in infective endocarditis study (ENDOVAL 1), the first randomized in endocarditis, will provide crucial information regarding the putative benefit of early surgery over the state-of-the-art therapeutic approach in high-risk patients with infective endocarditis.

DETAILED DESCRIPTION:
BACKGROUND Whereas mortality has been dramatically reduced in some areas of cardiac diseases thanks to continuous progress in treatment, endocarditis remains a high-mortality disease with steady percentages of mortality in the last 30 years. Several reasons may help to account for this frustrating comparison. The changing pattern of the epidemiology of endocarditis surely has contributed to the still high mortality. Patients are older, prosthetic and nosocomial endocarditis are currently more frequent, and Staphylococcus aureus has increased as the causative agent. But clinical investigators on this field must be aware of our fault in not generating evidence-based investigations. A paucity of comprehensive information exists and high-quality evidence is lacking. In fact, not even a single randomized study is available regarding the most challenging decision in endocarditis which is to decide whether and when surgery has to be undertaken in the active phase of the disease. Therefore, guidelines on treatment in endocarditis endorsed by the most prestigious scientific societies are supported by moderate (level B) or low level of evidence (level C). Not even a single recommendation on medical versus surgical treatment is based on a high level of evidence (level A). Unfortunately, it is still true that "there is still as much art as science in the care of patients with endocarditis". The only way investigators can balance the tip in favour of science is promoting randomized clinical studies with power enough to answer unsettled crucial clinical questions. Some encourage taking this track; it has been suggested by others, however, that a randomized study comparing medical versus surgical treatment in endocarditis cannot be undertaken.

American and European guidelines state with level of evidence B or C, and with subtle differences, that surgery should be considered in active endocarditis in the following situations: heart failure, valve abnormalities (dehiscence, perforation or rupture), periannular complications, persistent vegetation after systemic embolization, increase in vegetation size despite appropriate antibiotics, persistent infection, and infection by microorganisms known not to be cured by antimicrobial therapy.

All those indications are well-known predictors of poor short-term outcome in infective endocarditis and surgery is presumed to favourably alter that prognosis. However, it is already known that results of surgery are worse if patients have heart failure or persistent infection. Besides, those predictors very frequently appear after several days after the initial diagnosis. Finally, early surgery in active endocarditis has shown a lower mortality when compared to the usual medico-surgical approach. Based on this background, we hypothesize that if we wait for predictors of poor prognosis to appear, surgery may come too late. If, nonetheless, surgery is performed within the first 3 days after admission in patients with a high-risk profile before the clinical course worsens, prognosis may be improved. To test this hypothesis, factors which define early high-risk profile have to be identified. With this aim, we undertook a prospective, multicenter study in 317 patients with left-sided endocarditis and demonstrated that heart failure, Staphylococcus aureus and periannular complications detected within 72 hours after admission identified patients with poor prognosis.

In summary, predictors of poor prognosis available within 72 hours after admission can accurately identify high-risk patients. The initial clinical profile and the results of the first transesophageal echocardiogram and the initial blood cultures are accurate enough to stratify patients into high- and low-risk. Whether early surgery can improve prognosis when undertaken in the former is an attractive hypothesis never tested so far.

Once we are able to early identify a high-risk profile in infective endocarditis the following step has to be a randomized study in which the state-of-the-art therapeutic strategy for patients with endocarditis (medical treatment and surgery if predictors of poor prognosis appear early or late in the disease process) is compared to an early surgical approach. Of course, surgery and medical treatment cannot be compared and it would unethical doing so. What we are designing is a study to compare two different therapeutical strategies in high-risk patients, the state-of-the art approach, proposed by the international societies, and the early surgery strategy which includes two consecutive steps: 1) identification of high-risk patients by means of predictors available within 72 hours of admission; 2) surgery within 48 hours of inclusion of a patient in the high-risk group.

METHODS

Study hypothesis Our hypothesis is that early surgery in high-risk patients with active infective endocarditis decreases mortality and should be considered the treatment of choice in this population.

Study objectives Our objective is to compare the 30 days mortality rate in high-risk patients with active infective endocarditis between an early surgical approach (surgery performed within the first 48 hours after inclusion or 5 days after the initial diagnosis) and the state-of-the-art treatment in this disease (medical treatment followed by surgery if predictors of poor prognosis appear early or late).

Study population Our initial study population is made up of patients with active infective endocarditis in the initial phase of the disease (less than 5 days of the diagnosis) who do not meet the exclusion criteria (table I). Diagnosis of infective endocarditis will be performed according to modified Duke criteria. Patients who require urgent surgery (heart failure, septic shock, or fungal endocarditis) are rapidly sent to surgery. Patients with more than 5 days between the diagnosis and the first contact with our centres are excluded since the concept of early surgery cannot be applied to them. A surgical risk over 40% calculated by means of the logistic Euroscore system are also excluded since their preoperative status is so poor that the surgical risk prohibits a surgical approach. Patients with ischemic or hemorrhagic stroke are also excluded given its very difficult management during the perioperative period which may introduce bias in the results.

Study design Patients without any exclusion criteria will be divided into two groups according to the risk profile. When the patient does not fulfil any of the high-risk criteria, he or she is considered a low-risk patient and is managed with the state-of-the-art therapeutic strategy, according to the guidelines accepted by the different international societies: medical management by a multidisciplinary team is accomplished. A complete clinical examination is done every day. Blood and urine analysis, chest X-ray, EKG and blood cultures are taken initially, and every 7 days. Transthoracic and ransesophageal echocardiography is performed initially. All the previous tests, including transesophageal echocardiography, are performed always the clinical status changes. CT scan is indicated when stroke or peripheral emboli are clinically suspected. Surgery is considered and decided in an individual basis when any of the following is present: heart failure, periannular complications, persistent >10 mm vegetation after systemic embolization, or persistent infection (fever or positive blood cultures after 7 days of correct antibiotic treatment once other sources of fever are ruled out). The specific surgical technique will be decided by the surgeon according to the degree of tissular destruction and will be aimed to remove the infected tissue and to repair the damaged structures or, if this is not feasible, to implant cardiovascular prosthesis.

If the patient meets any of the high-risk criteria, he or she is randomized to the state-of-the-art therapeutic strategy aforementioned or the early surgical strategy. In the latter, surgery must be performed within 48 hours after randomization. Therefore, the time from the first contact to the hospital to surgery cannot be longer than 5 days (3 days to have the transesophageal exam and the blood cultures available and 2 days for randomization to surgery). The study flow chart is shown in figure 1.

The only event to be considered in the statistical analysis will be death within 30 days of admission. The study will be prolonged and patients will be followed for 1 year. In the long-term analysis death and a new episode of endocarditis will be considered the only events. Table II depicts the study schedule and procedures. Table III depicts the long-term substudy schedule and procedures

The protocol has been approved by the local ethical committee of the following institutions: 1) Universitary Clinic Hospital, Valladolid, Spain; 2) Universitary Clinic Hospital San Carlos, Madrid, Spain; 3) Universitary Clinic Hospital Valle Hebrón, Barcelona, Spain. It is currently being evaluated by cardiologists and cardiac surgeons from: 1) Universitary Clinic Hospital Gregorio Marañón, Madrid, Spain; 2) Clínic Hospital, Barcelona, Spain; 3) German Trias i Pujol Hospital, Badalona, Barcelona, Spain.

STATISTICAL CONSIDERATIONS Determination of sample size The study will be powered to address the primary hypothesis that a decision to operate on an urgent basis patients with high-risk endocarditis will decrease in-hospital mortality compared to patients managed with the state-to-art strategy. Thus, the sample size was calculated based on the assumption of an 30% of mortality in the state-to-art group (19) versus 13% in the early surgery group (17% relative reduction). A sample size of 206 patients will produce a study power of 80% with a 2-sided α level of .05. As a result, assuming a 5% of losses during the study period, a sample size of 216 enrolled patients is needed with 108 in each group.

Randomization Once the patient has complied with protocol requirements and has signed the informed consent, he or she will be included in the study and randomized to one of the two strategies. Randomization will be performed with blocks of four and six patients by an automated assignment system. Blocks will be re-randomized to avoid knowing block size. All calculations have been performed with C4-Study design pack (Glaxo Wellcome V1.1)

The independence will be guaranteed because the person who makes the process will be contact by telephone and will not take any clinical decision about the patient.

Safety issues An intermediate analysis will be done to control the quality of the information collected and to contrast the hypothesis of the study. The study will be stopped if a rate of adverse event higher than expected is observed.

Statistical analysis Once that information has been collected and checked, the statistical analysis will begin. Statistical analysis of data will follow the intention-to-treat principle, that is, patients will be analyzed according to the treatment arm to which they were randomized, regardless of adherence to the assigned treatment. Continuous variables will be compared with t-Student test and U Mann-Whitney test for non-normally distributed variables and categorical variables will be compared with Chi-Square test and Fisher's exact test when appropriate.

The distribution of time to event variables will be estimated by the Kaplan-Meier method, treatment effects will be compared with log-rank test. The Cox regression method will be used to estimate the hazard ratio and 95% confidence interval. All test will be two-sided and p values of less then 0.05 will be considered to indicate statistical significance. Statistical analysis will be performed with SPSS software V 14.0 (SPSS Inc., Chicago, IL, USA)

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Infective endocarditis diagnosed by modified Duke criteria.
* At least one of the following risk factors:

  1. Periannular complications
  2. New onset auriculo-ventricular block
  3. New onset severe valvular insufficiency
  4. Early-onset prosthetic valve endocarditis
  5. Staphylococcus aureus endocarditis
  6. Vegetations greater than 20 mm

Exclusion Criteria:

* Patients with urgent/emergent indication of surgery when endocarditis is diagnosed:

  1. Heart failure because of valvular insufficiency.
  2. Fungal endocarditis.
  3. Septic shock.
* Patients referred from other centers to be operated on.
* Patients without echocardiographic evidence of endocarditis.
* Pregnant or lactating women.
* Simultaneous participation in other research study.
* Incapacity to mantein the conditions of the study.
* Patients referred from other centers more than 5 days after the diagnosis of infective endocarditis.
* Patients with prohibitive risk for surgery due to comorbidities, estimated by previous validated scales. An Euroescore value greater than 40% will be considered a contraindication to enter the protocol.
* Patients with ischemic or haemorragic stroke within one month before the diagnosis of endocarditis.
* Endocarditis in intravenous drug addicts patients.
* Not signed the inform consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2007-09; Primary Completion 2007-11 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality rate in high-risk patients with active infective endocarditis between an early surgical approach and the state-of-the-art treatment in this disease. | In-hospital mortality

SECONDARY OUTCOMES:
One year mortality rate in high-risk patients with active infective endocarditis between an early surgical approach and the state-of-the-art treatment in this disease. | One year

CONTACTS AND LOCATIONS:
Overall Officials: José A San Román, MD, FESC, Principal Investigator — Instituto de Ciencias del Corazon
Locations (1):
- Universitary Hospital of Valladolid, Valladolid, Spain

REFERENCES:
- [Derived] Fernandez-Hidalgo N, Almirante B, Tornos P, Gonzalez-Alujas MT, Planes AM, Larrosa MN, Sambola A, Igual A, Pahissa A. Prognosis of left-sided infective endocarditis in patients transferred to a tertiary-care hospital--prospective analysis of referral bias and influence of inadequate antimicrobial treatment. Clin Microbiol Infect. 2011 May;17(5):769-75. doi: 10.1111/j.1469-0691.2010.03314.x. PMID 20636419
- [Derived] San Roman JA, Lopez J, Revilla A, Vilacosta I, Tornos P, Almirante B, Mota P, Villacorta E, Sevilla T, Gomez I, Del Carmen Manzano M, Fulquet E, Rodriguez E, Igual A. Rationale, design, and methods for the early surgery in infective endocarditis study (ENDOVAL 1): a multicenter, prospective, randomized trial comparing the state-of-the-art therapeutic strategy versus early surgery strategy in infective endocarditis. Am Heart J. 2008 Sep;156(3):431-6. doi: 10.1016/j.ahj.2008.04.006. Epub 2008 Jul 2. PMID 18760122